CLINICAL TRIAL: NCT05058300
Title: Prospective Registry for Patients With Chest Pain in Emergency Department
Acronym: ThReg
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jena University Hospital (Other)
Collaborators: Zentrum für Klinische Studien Jena (Other); GE Healthcare (Industry)
Responsible Party: Principal Investigator, Ulf Teichgräber, Prof. Dr. med., Jena University Hospital
Other Study IDs: 5149-04/17
Record Dates: First submitted 2017-07-17; First posted 2021-09-27 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Chest Pain
Keywords: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Chest Pain: An unselected patient-population with chest pain in emergency department
  Interventions: Device: CT Thorax

INTERVENTIONS:
Device: CT Thorax — CT Thorax (GE Revolution with chest pain algorithm)

SUMMARY:
monocentric, prospective registry collection of clinical data of all patients with chest pain in emergency department and follow-up after 30 days

DETAILED DESCRIPTION:
An unselected patient-population with chest pain entering through the emergency department participate in a diagnostic survey where a chest pain algorithm based mainly on risk scores (Grace, TIMI, Heart) verifying the diagnostic forecasting power (sensitivity, specificity, negative and positive predictive value) of biomarkers, risk scores and imaging methods for diagnosing of potential life-threatening disease.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old chest pain written confirmation of participants or legal representative

Exclusion Criteria:

* thorax trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An unselected patient-population with chest pain in emergency department
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2024-10-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic forecast of biomarkers, risk scores and computer tomography | From admission to emergency unit discharge
  Diagnostic forecast compared to the initial suspected diagnosis and discharge diagnosis

SECONDARY OUTCOMES:
Sensitivity | During diagnostic procedure
  Sensitivity in result of biomarkers, risk scores and imaging methods
Specificity | During diagnostic procedure
  Specificity in result of biomarkers, risk scores and imaging methods
Positive predictive value | During diagnostic procedure
  Positive predictive value in result of biomarkers, risk scores and imaging methods
Negative predictive value | During diagnostic procedure
  Negative predictive value in result of biomarkers, risk scores and imaging methods
Major adverse cardiac events (MACE) | From admission to emergency unit until 30 days after or death
  outcome is measured by coronary intervention, coronary bypass and death within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Behringer, Prof., Principal Investigator — Emergency Unit, University hospital Jena
Locations (1):
- Department of Emergency, Jena, Thuringia, Germany